CLINICAL TRIAL: NCT02515565
Title: Effects of a Physiotherapy Program in Patients Hospitalized Due to Pneumonia
Brief Title: Physiotherapy in Patients Hospitalized Due to Pneumonia.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, PhD, Universidad de Granada
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: DF0057UG
Record Dates: First submitted 2015-08-02; First posted 2015-08-04 (Estimated); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Pneumonia
Keywords: pneumonia; Exacerbation; physiotherapy; hospitalization
MeSH Terms: conditions — Pneumonia | interventions — Cephalosporins; Erythromycin; Physical Therapy Modalities; Transcutaneous Electric Nerve Stimulation; Breathing Exercises

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental group (Experimental): Patients with a clinical diagnosis of pneumonia will be included in this group. They will be included in a physiotherapy program added to the standard medical treatment.
  Interventions: Other: Physiotherapy program
- Control group (Other): Patients with a clinical diagnosis of pneumonia will be included in this group. They will receive only the standard medical treatment based on cephalosporin with or without erythromycin.
  Interventions: Drug: cephalosporin with or without erythromycin

INTERVENTIONS:
Drug: cephalosporin with or without erythromycin — Second- or third-generation cephalosporin (cefuroxime, cefotaxime, or ceftriaxone) with or without erythromycin, given parenterally; parenteral therapy should continue until the patient has been afebrile for more than 24 hours and oxygen saturation exceeds 95 percent.
  Other Names: Standard medical treatment
  Arms: Control group
Other: Physiotherapy program — The physiotherapy treatment will be performed during the hospitalization, every day during 45-60 minutes added to the standard medical treatment. I will include breathing exercises, electrostimulation in quadriceps with voluntary contraction and exercises with theraband.
  Other Names: Physiotherapy; Electrostimulation; Respiratory exercises
  Arms: Experimental group

SUMMARY:
Acute respiratory infections are the fourth cause of hospitalization in elderly. Various studies have examined the impact of hospitalization in patients with respiratory pathology, showing the need of interventions in order to reduce the impact of hospitalization. The objective of this study is to examine whether a physical therapy intervention can reduce impairment in patients hospitalized due to pneumonia.

DETAILED DESCRIPTION:
Acute respiratory infections are the fourth cause of hospitalization in elderly. Hospital admissions due to pneumonia range from the 1.1 and 4 per 1,000 patients, increasing with age. Hospitalization causes a decline in physical and functional status. Physical impairment involves a higher risk of disability and mortality in elderly people. Various studies have examined the impact of hospitalization in patients with respiratory pathology, and it has been shown that hospitalization implies a significant physical impairment in patients admitted for pneumonia showing that this deterioration increases with age. That highlights the need of interventions in order to reduce the impact of hospitalization. The objective of this study is to examine whether a physical therapy intervention can reduce impairment in patients hospitalized due to pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pneumonia.
* No contraindication of physiotherapy.
* Signed written consent.
* Medical approval for inclusion.

Exclusion Criteria:

* Contraindications of physiotherapy.
* Neurological, orthopedic or heart disease.
* Prosthetic devices in lower limbs.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Muscle strength | Participants will be followed for the duration of hospital stay, an expected average of 8 days
  Quadriceps strength will be assessed with a portable dynamometer. The test will be performed as previously reported.
Exercise capacity | Participants will be followed for the duration of hospital stay, an expected average of 8 days
  Five times sit to stand test (5STS) will be used to assess exercise capacity, 5STS is a simple assessment tool that is feasible in all healthcare settings, and may be a rapid method of assessing changes in exercise capacity in COPD and screening for poor physical functioning individuals.

SECONDARY OUTCOMES:
Respiratory function | Participants will be followed for the duration of hospital stay, an expected average of 8 days
  Spirometry is regarded as the gold standard measure of respiratory function. Spirometry will be performed according to the American Thoracic Society (ATS) criteria.
Dyspnea perception | Participants will be followed for the duration of hospital stay, an expected average of 8 days
  Dyspnea perception will be assessed with Borg modified scale. Patients will classify their breathlessness between 0 and 10.
Quality of life | Participants will be followed for the duration of hospital stay, an expected average of 8 days.
  EuroQol-5D (EQ-5D) will be used to assess quality of life. EQ-5D is a generic questionnaire and consists of two parts, the EQ-5D Visual analogue scale (VAS) and the EQ-5D index. The EQ-5D VAS consists on a vertical rating scale from 0 to 100 (0 = death/worst possible health state and 100 = best possible health state). The EQ-5D index is a five-item questionnaire (mobility, self-care, usual activity, pain/discomfort and anxiety/depression). Each item has three levels: no problem, some problem and severe problem.
Functionality | Participants will be followed for the duration of hospital stay, an expected average of 8 days.
  The London Chest Activity of Daily Living (LCADL) is a valid tool that is validated to measure breathlessness during daily activities. It is a 15-item questionnaire divided in 4 domains: self-care (4 items), domestic (6 items) physical activity (2 items) and leisure (3 items).
Fatigue | Participants will be followed for the duration of hospital stay, an expected average of 8 days.
  Fatigue will be assessed with the Fatigue Severity Scale (FSS). The FSS is a nine-item instrument designed to assess fatigue as a symptom of a variety of different chronic conditions and disorders. The scale addresses fatigue's effects on daily functioning, querying its relationship to motivation, physical activity, work, family, and social life, and asking respondents to rate the ease with which they are fatigued and the degree to which the symptom poses a problem for them.
Mood | Participants will be followed for the duration of hospital stay, an expected average of 8 days.
  Mood in these patients will be measured by the Hospital Anxiety and Depression Scale.

OTHER OUTCOMES:
Dependency levels | Baseline
  Dependency levels will be evaluated with the Functional Independence Measure (FIM). It is an 18-item, 7-level scale developed to uniformly assess severity of patient disability and medical rehabilitation functional outcome.
Comorbidities | Baseline
  Charlson Comorbidity Index will be used to assess the comorbidities of the patients, it is a simple and valid method of estimating risk of death from comorbid disease. It contains 19 categories of comorbidity and predicts the ten-year mortality for a patient who may have a range of co-morbid conditions. Each condition is assigned with a score of 1, 2, 3 or 6 depending on the risk of dying associated with this condition.
Nutritional status | Baseline
  Nutritional status was evaluated with Mini nutritional assessment (MNA) test, that is validated to provide a single, rapid assessment of nutritional status in elderly patients in outpatient clinics, hospitals, and nursing homes. The MNA test is composed of simple measurements and brief questions that can be completed in about 10 min.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Carmen Valenza, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Faculty of Health Sciences. University of Granada., Granada, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lopez-Lopez L, Torres-Sanchez I, Rodriguez-Torres J, Cabrera-Martos I, Ortiz-Rubio A, Valenza MC. Does adding an integrated physical therapy and neuromuscular electrical stimulation therapy to standard rehabilitation improve functional outcome in elderly patients with pneumonia? A randomised controlled trial. Clin Rehabil. 2019 Nov;33(11):1757-1766. doi: 10.1177/0269215519859930. Epub 2019 Jun 27. PMID 31244327